CLINICAL TRIAL: NCT00085306
Title: Phase II Trial Of Interferon-B In Patients With Metastatic Cutaneous Melanoma And Metastatic Ocular Melanoma
Brief Title: Interferon Beta in Treating Patients With Metastatic Cutaneous Melanoma or Ocular Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE1604; P30CA043703 (NIH); CCF-4049 (Other: Cleveland Clinic IRB); CASE1604 (Other: Case Comprehensive Cancer Center)
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-10

CONDITIONS: Stage IV Melanoma; Recurrent Melanoma
Keywords: recurrent melanoma; stage IV melanoma; iris melanoma; ciliary body and choroid melanoma, medium/large size; extraocular extension melanoma; recurrent intraocular melanoma
MeSH Terms: conditions — Melanoma; Uveal Melanoma | interventions — Interferon-beta

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Recombinant interferon beta (Experimental)
  Interventions: Biological: recombinant interferon beta

INTERVENTIONS:
Biological: recombinant interferon beta — recombinant interferon beta

SUMMARY:
RATIONALE: Interferon beta may interfere with the growth of tumor cells.

PURPOSE: This phase II trial is studying how well interferon beta works in treating patients with metastatic cutaneous (skin) melanoma or ocular (eye) melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the objective clinical response rate in patients with metastatic cutaneous or ocular melanoma treated with interferon beta.
* Determine the frequency and degree of apoptosis induction in patients treated with this drug.
* Determine the safety and tolerability of this drug in these patients.

OUTLINE: This is an open-label study. Patients are stratified according to type of melanoma (ocular vs cutaneous).

Patients receive interferon beta subcutaneously once daily in the absence of disease progression or unacceptable toxicity.

Patients are followed within 3 days after completion of study treatment and then for survival.

PROJECTED ACCRUAL: A total of 28-56 patients (14-28 per stratum) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic melanoma

  * Cutaneous or ocular disease
* Measurable disease
* No active unstable CNS metastases by neurologic exam AND CT scan or MRI

  * Irradiated and/or resected CNS lesions allowed if there is no evidence of disease by head MRI or CT scan for > 6 months after surgery and/or radiotherapy
  * Patients with cutaneous metastases and previously irradiated and/or resected CNS metastases are eligible if the CNS metastases are controlled and do not require dexamethasone

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1 (0-2 for patients with cutaneous metastases)

Life expectancy

* At least 3 months

Hematopoietic

* Absolute neutrophil count ≥ 1,200/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9.5 g/dL

Hepatic

* Bilirubin ≤ 1.5 mg/dL
* AST ≤ 3.0 times normal
* Alkaline phosphatase ≤ 2.5 times normal (10 times normal if due to bone metastases)
* Hepatitis B surface antigen negative

Renal

* Creatinine ≤ 1.5 mg/dL

Cardiovascular

* No serious cardiac arrhythmia requiring treatment
* No congestive heart failure
* No angina pectoris
* No New York Heart Association class II-IV heart disease
* No other severe cardiovascular disease

Other

* HIV negative
* No other malignancy within the past 3 years except basal cell or squamous cell skin cancer or carcinoma in situ of the uterine cervix
* No history of seizure disorder
* No severe psychiatric disorder
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 12 months since prior adjuvant interferon alfa-2 (IFNα-2) therapy
* More than 30 days since prior IFNα-2 therapy for metastatic disease (6 months for patients with cutaneous metastases)
* No more than 1 prior systemic regimen (chemotherapy or biologic) for metastatic disease (3 regimens for patients with cutaneous metastases)

Chemotherapy

* See Biologic therapy
* No concurrent chemotherapy

Endocrine therapy

* See Disease Characteristics
* Concurrent replacement therapy with physiologic doses of corticosteroids allowed

  * No concurrent dexamethasone or other steroidal antiemetics or anti-inflammatories
* No other concurrent hormonal agents except steroids administered for preexisting adrenal failure or hormones administered for non-disease-related conditions (e.g., insulin for diabetes)

Radiotherapy

* See Disease Characteristics
* More than 28 days since prior radiotherapy and recovered
* No concurrent palliative radiotherapy

Surgery

* See Disease Characteristics
* No prior organ allograft
* More than 28 days since prior major surgery requiring general anesthesia

Other

* More than 28 days since prior antibiotics for local or systemic infection
* No concurrent aspirin
* No concurrent barbiturates
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2004-04; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Objective clinical response rate to IFN-B the maximum tolerated dose as measured by a CTC Grade III hematologic or a Grade IV granulocyte toxicity which persists > 3 days at 1 week after each course

CONTACTS AND LOCATIONS:
Overall Officials: Ernest C. Borden, MD, Study Chair — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States